CLINICAL TRIAL: NCT03831958
Title: Long-Term Follow-UP of Survivors of Pediatric Cushing Disease
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190051; 19-CH-0051
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10-01

CONDITIONS: Cushing Disease
Keywords: Body Mass Index Z Score; Adult Height; Endocrine Function; Neuropsychological Outcome; Metabolic Syndrome; Natural History
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family member: Family member of survivor of pediatric Cushing disease
- Subjects: survivor of pediatric Cushing disease

SUMMARY:
Background:

The pituitary gland produces hormones. A tumor in this gland can cause it to produce too much of the hormone cortisol. Too much cortisol in the body causes Cushing disease. This disease causes many problems. Some of these problems might persist after the disease is cured.

Objective:

To find out the long-term effects of exposure to high levels of cortisol during childhood and adolescence.

Eligibility:

People ages 10-42years who were diagnosed with Cushing disease before age 21 and are now cured and have normal or low cortisol levels

People related to someone with Cushing disease

Design:

Participants will be screened with a medical history.

Participants will complete an online survey. This will include questions about their or their child s physical and mental health.

All participants will be seen at 5 -year intervals after cure of Cushing disease (5yr, 10yr, 15yr, 20yr (last visit))

Participants who have a relative with Cushing disease will have a medical history and blood tests or cheek swabs.

Participants who have the disease will have:

Physical exam

Blood tests

Cheek swab

DXA scan: A machine will x-ray the participant s body to measure bone mineral content.

For participants who are still growing, a hand x-ray

Participants with the disease may also have:

Hormone stimulation test: Participants will get a hormone or another substance that will be measured.

Serial hormone sampling: Participants blood will be measured several times through a thin plastic tube in an arm vein.

Urine tests: Participants urine may be collected over 24 hours.

MRI: Participants may have a dye injected into a vein. They will lie on a table that slides into a machine. The machine will take pictures of the body.

DETAILED DESCRIPTION:
Objective:

Cushing Disease (CD) describes the state of hypercortisolemia secondary to cortisol producing pituitary adenomas. The rarity of the disease (2-5 new cases per million, 1 out of 10 in children) and the subtle initial findings result in prolonged undiagnosed hypercortisolemia, that increases the risk for significant complications, including obesity, height deceleration, hyperlipidemia, hyperglycemia, hypertension, osteoporosis, immunodeficiency, and others. Although hypercortisolemia usually resolves after successful resection of the pituitary adenoma, the reversal of the abovementioned complications and the long-term effects of the previous prolonged exposure of the body to supraphysiologic levels of cortisol have not been clarified, especially when hypercortisolemia occurs during childhood.

Previous studies have addressed the possible complications after resolution of hypercortisolemia, but most of them refer to adult patients. Amongst the described complications, suppression of the pituitary hormones, such as the growth and thyroid hormone axes, and persistent increase of the body mass index (BMI) and abnormal fat distribution, have been described in limited number of pediatric patients followed for a few years after cure. Other complications, such as components of the metabolic syndrome or cardiovascular dysfunction, have not been extensively studied in children. Furthermore, equally important are the long-term effects of glucocorticoids on other aspects of health. For example, it has been previously described that the neurocognitive function of children with CD declines the first year after treatment. This can potentially result in impaired quality of life, lower education level, and lower job and life satisfaction in the future; however, the long-term neurocognitive sequelae of Cushing syndrome (CS) diagnosed in childhood have not been studied.

This study aims to provide novel insight on the long-term effects of hypercortisolemia on the developing child, their underlying pathogenetic mechanisms, their evolution over time, and the risk factors for developing them. This will assist in designing methods to closely monitor or prevent them in the future. Certain results of this study could potentially apply to children with iatrogenic CS, which is much more common due to the widespread use of pharmacologic doses of glucocorticoids in malignancies, autoimmune and atopic disorders.

Study population:

The study population will consist of patients that were previously successfully treated for CD before the age of 21 years. We aim to identify these patients through review of our current protocol 97-CH-0076 on "Clinical and genetic investigation of pituitary and hypothalamic tumors", which has been recruiting patients since 1997. We will also accept patients who have been diagnosed and successfully treated for pediatric CD at outside institutions after reviewing the medical records and confirming their diagnosis. The patients must not be hypercortisolemic at the time of their recruitment. Family members (any age) of patients with a family history of pituitary tumors and who will agree to participate in the DNA/linkage analysis study.

Design:

We will evaluate patients at specific intervals after cure at 5 (+/-1), 10 (+/-1), 15 (+/-1) and 20 (+/-1) years after documented resolution of hypercortisolemia.

The study will include an online survey offered to all patients, as well as an on-site short visit for those willing to travel to NIH.

The online survey will include questionnaires on assessment of various aspects of health: Current medical diagnoses, Medication use, History of endocrine disorders, Fertility, Quality of life, Behavioral and emotional symptomology, and Socioeconomic and Demographic information. The survey will be developed and distributed with the help of CTDB and will be sent with secure email to all the patients and/or their parents (for patients who are <18yo at the time of evaluation) after consent and eligibility have been confirmed.

The short on-site visit at NIH will be offered to all the patients willing to travel. Blood tests, imaging studies (MRI pituitary/brain and DXA scan), and neurocognitive screening and patient reported outcome questionnaires will be performed.

Outcome measures:

The primary outcome measure of the study is the difference of the Body Mass Index (BMI) z-score of the patients previously treated for pediatric CD compared to the general population, as calculated by data derived from the NHANES study.

The secondary outcomes will be to describe the prevalence of other endocrine and non-endocrine abnormalities after successful treatment of CD in childhood, including: growth hormone, thyroid, gonadal, adrenal function; bone mineral density; glucose metabolism; lipid profile; cardiovascular abnormalities; immunologic changes; coagulation function; psychiatric diseases, behavioral symptomology; neurocognitive function; and quality of life.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females 10-42 years old (subjects) who were previously diagnosed and had successful treatment of CD before the age of 21 years old. Patients who have undergone therapies other than surgical resection (such as radiation or medical treatment) will be eligible to participate.
  2. Normocortisolemia or hypocortisolemia at the time of the study (as documented within past 6 months of recruitment) documented as urine free cortisol or midnight/afternoon serum or salivary cortisol levels within or below the normal range or documented panhypopituitarism (on glucocorticoid replacement).
  3. Patients or a legal guardian (in case of cognitively impaired adults or children) must provide assent/consent at the time of the recruitment.
  4. Family members (2- 90 yrs.) of patients with a family history of pituitary tumors and who agree to participate in the DNA/linkage analysis study.

EXCLUSION CRITERIA:

1. Pregnancy
2. Patients with any medical, physical, psychiatric, or social conditions, which, in the opinion of the investigators, would make participation in this protocol not in their best interest, will be excluded from the on-site visit of the study. Patients who are critically ill, unstable, or with severe organ failure that may affect/limit the endocrine evaluation and place unsustainable demands on Clinical Center or NICHD resources will be excluded. They will still be offered the opportunity to participate in the online questionnaire part of the study.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients that were previously successfully treated for CD before the age of 21 years. We aim to identify these patients through review of our current protocol 97-CH-0076 on Clinical and genetic investigation of pituitary and hypothalamic tumors , which has been recruiting patients since 1997. We will also accept patients who have been diagnosed and successfully treated for pediatric CD at outside institutions after reviewing the medical records and confirming their diagnosis. The patients must be normocortisolemic at the time of their recruitment. Family members of subjects who are survivors of pediatric Cushing disease will be invited to participate in the DNA/linkage analysis study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2040-01-03 (Estimated); Study Completion 2040-01-03 (Estimated)

PRIMARY OUTCOMES:
Difference in body mass index z-score of subjects previously treated for Cushing disease compared to general population | baseline, 5, 10, 15, 20 years
  The primary outcome measure of the study is the difference in the Body Mass Index (BMI) z-score of the patients previously treated for pediatric CD compared to the general population, as calculated by data derived from the NHANES study.

SECONDARY OUTCOMES:
Prevalence of endocrine and non-endocrine abnormalities | baseline, 5, 10, 15, 20 years
  The secondary outcomes will be to describe the prevalence of other endocrine and non-endocrine abnormalities after successful treatment of CD in childhood, including: growth hormone, thyroid, gonadal, adrenal function; bone mineral density; glucose metabolism; lipid profile; cardiovascular abnormalities; immunologic changes; coagulation function; psychiatric diseases, behavioral symptomology; neurocognitive function; and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stratakis CA. Diagnosis and Clinical Genetics of Cushing Syndrome in Pediatrics. Endocrinol Metab Clin North Am. 2016 Jun;45(2):311-28. doi: 10.1016/j.ecl.2016.01.006. PMID 27241967
- [Background] Davies JH, Storr HL, Davies K, Monson JP, Besser GM, Afshar F, Plowman PN, Grossman AB, Savage MO. Final adult height and body mass index after cure of paediatric Cushing's disease. Clin Endocrinol (Oxf). 2005 Apr;62(4):466-72. doi: 10.1111/j.1365-2265.2005.02244.x. PMID 15807878
- [Background] Keil MF, Graf J, Gokarn N, Stratakis CA. Anthropometric measures and fasting insulin levels in children before and after cure of Cushing syndrome. Clin Nutr. 2012 Jun;31(3):359-63. doi: 10.1016/j.clnu.2011.11.007. Epub 2011 Dec 7. PMID 22154461
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-CH-0051.html